CLINICAL TRIAL: NCT01173172
Title: A Phase I/II Trial of Boron Neutron Capture Therapy (BNCT) for Recurrent Head and Neck Cancer at Tsing-Hua Open Pool Reactor
Brief Title: Boron Neutron Capture Therapy (BNCT) for Locally Recurrent Head and Neck Cancer
Acronym: BNCT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Tsing Hua University,Taiwan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BNCT_090514
Record Dates: First submitted 2010-07-28; First posted 2010-07-30 (Estimated); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Head and Neck Cancer
Keywords: Boron neutron capture therapy (BNCT); Head and neck cancer; toxicities; response rate
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Boron Neutron Capture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BNCT, recurrent head and neck cancer (Experimental): Single arm treated by BNCT only
  Interventions: Radiation: Boron Neutron Capture Therapy

INTERVENTIONS:
Radiation: Boron Neutron Capture Therapy — Boronophenylalanine (BPA) 500 mg/kg on D1 and D30 followed by BNCT for 2 fractions (D1 and D30)

SUMMARY:
This is a boron neutron capture (BNCT) therapy for patients with previously irradiated and locally recurrent head and neck cancer. The primary end points are treatment toxicities and response rate. The secondary endpoints are time to tumor progression, progression-free survival, overall survival and change quality of life.

Head and neck carcinomas that recur locally after conventional irradiation pose a therapeutic challenge. Boron neutron capture therapy (BNCT) is based on the nuclear capture reaction that occurs when non-radioactive boron is irradiated with neutrons of thermal energy to yield high energy alpha particles and recoiling lithium nuclei. The effect of alpha and 7Li is primarily limited to boron- containing cells. Preferential uptake of boron into cancerous tissue is achieved using boron carriers such as a derivative of phenylalanine, boronophenylalanine (BPA). After administration of BPA by an intra-arterial or intravenous infusion, the tumor site is irradiated with neutrons, the source of which is currently a nuclear reactor. A few uncontrolled clinical trials have evaluated BNCT in the treatment of glioblastoma after brain surgery. In these studies, the median survival times have been 13-15 months after BNCT. However, efficacy and tolerability of BNCT in the treatment of limited number of head and neck cancer patients showed promising results. Though many basic researches about BNCT has been done using Tsing Hua Open-pool Reactor (THOR) at National Tsing Hua University, no clinical trial utilizing BNCT is performed in our country. This study will be the first BNCT trial to treat head and neck cancer in Taiwan.

DETAILED DESCRIPTION:
This is a prospective, single arm, open label phase I/II trial with boron neutron capture (BNCT) therapy for patients with previously irradiated and locally recurrent head and neck cancer.

The eligibility criteria are patients with locoregionally recurrent head and neck cancer; good performance status; inoperable, clinical measurable tumor size; good organ function and good compliance. No systemic treatment is in use. Once entering this study, patients will receive angiographies to evaluate bloody supply of the tumor and PET scan with 18F-fluoro-L-BPA as the tracer. Tumor-to- normal tissue ratios were evaluated from static emission scans. Boron concentration of normal tissues is derived from measurement of BPA concentration in the blood. Treatment planning with THORplan will be done after Computerized Tomography (CT) simulation. After treatment plan approved and on the day of treatment, intravenous or intra-arterial L-BPA- Fructose complex 500 mg/kg was administered at a constant rate over about 3 hours before and during neutron irradiation. Neutron beam irradiations were given at the THOR with prescription dose of 20 to 25 Gy (Eq) for the tumor in one fraction on day 1 and repeated on day 30. Patients will be regularly followed up at OPD for toxicities (NCI Common Terminology Criteria) and response evaluation (RECIST criteria)by MRI and PET, time to progression measurement, survival status and change of quality of life. Maximally 27 patients will be enrolled. After first 10 patients, the preliminary results will be reviewed before further patients' enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locoregionally recurrent, histologically proved malignancy of the head and neck.
* Prior conventional radiotherapy administered has been given for the disease (except melanoma) and surgery, conventional radiotherapy or chemotherapy are not appropriate for salvage.
* Bi-dimensionally measurable disease by MRI and/or CT scan and ≦ 12 cm in largest dimension.
* Age greater than 18 years and < 80 years, ECOG performance status ≦ 2
* WBC > 2.5 x109/L, neutrophil count >1.0 x109/L, platelet count >75x109/L, serum creatinine <1.25xULN.
* Informed consent signed.
* Tumor to Normal tissue (T/N) ratio for BPA >2.5 by 18F-BPA PET scan.

Exclusion Criteria:

* Lymphoma or other tumor type that is expected to respond to cancer chemotherapy or to a dose of conventional radiation therapy that can be safely given.
* Patients who had an effective standard treatment option available.
* Distant metastasis outside of the head and neck region.
* Expecting life less than 3 months.
* A time interval less than 3 months from previous radiation therapy.
* Concurrent systemic cancer treatment including chemotherapy or target therapy.
* Severe congestive heart failure or renal failure.
* Pregnancy.
* Restless patients who were unable to lie or sit in a cast for 30-60 min.
* A cardiac pace-maker or an unremovable metal implant present in the head and neck region that will interfere with MRI-based dose-planning or tumor response evaluation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2014-03-07 (Actual); Study Completion 2015-03-07 (Actual)

PRIMARY OUTCOMES:
Treatment toxicities and response rate | 2 years
  CTC ver 4 for toxicities RECIST for response

SECONDARY OUTCOMES:
Time to tumor progression | 5 year
  Interval between enrollment to disease progression
Progression-free survival | 5 years
  Percentage of patients without any disease progression at a time point
overall survival | 5 year
  Percentage of surviving patients at a time point
Change of quality of life | 2 year
  Health-related quality of life will be measured before and after BNCT at regular intervals

CONTACTS AND LOCATIONS:
Overall Officials: Ling-Wei Wang, MD, Principal Investigator — Cancer Center, Veterans General Hospital-Taipei, Taiwan
Locations (1):
- Cancer Center, Taipei Veterans General Hospital, Taipei, Taiwan